CLINICAL TRIAL: NCT06057766
Title: Physical Activity Coaching After Surgery for Patients With Resectable Non-small Cell Lung Cancer: a Randomized Controlled Trial
Brief Title: Physical Activity Coaching After Surgery for Patients With Resectable Non-small Cell Lung Cancer
Acronym: LucaMove
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Hasselt University (Other); AZ Sint-Jan AV (Other); AZ Delta (Other); Ziekenhuis Oost-Limburg (Other); Jessa Hospital (Other); KU Leuven (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONZ-2023-0153 - ID9994
Record Dates: First submitted 2023-06-22; First posted 2023-09-28 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer; Non-small Cell Carcinoma
Keywords: Surgery; Physical activity; coaching; telecoaching
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity tele coaching group (Experimental): Patients in the experimental group will undertake a 12-week (semi)automated telecoaching program with the aim of enhancing their physical activity. The program uses a Fitbit wearable and a smartphone application that is developed for and tested to be effective for patients with COPD.
  Interventions: Other: Physical activity tele coaching program
- Control group (No Intervention)

INTERVENTIONS:
Other: Physical activity tele coaching program — The program includes
  1. one-to-one semi-structured interview with the coach discussing the importance of physical activity, motivation, self-efficacy, barriers, favourite activities, and (coping) strategies to become more active resulting in an individual action plan;
  2. step counter (Fitbit) providing direct feedback which automatically sends data to the smartphone via blue-tooth. Patients will be asked to wear this step counter every day during the intervention;
  3. smartphone coaching application (mPAC), installed on a smartphone and linked to the step counter, will provide automated coaching by displaying an individual activity goal (expressed as daily step count) and daily and weekly feedback on the performance (steps) of the patient.
  4. phone calls by the coaches initiated in pre-defined situations (non-compliance with wearing the step counter, failure to transmit the data, failure to progress).
  Evidence-based behaviour change techniques will be implemented.
  Arms: Physical activity tele coaching group

SUMMARY:
The goal of this randomized controlled clinical trial is to test a 12-week physical activity telecoaching program for NSCLC patients after surgery.

The main question it aims to answer is:

What is the effectiveness and acceptability of a 12-week (semi)automated low-to-moderate intensity PA tele coaching program on physical activity (mean steps per day) in resectable (stage I-IIIA) NSCLC patients after lung surgery, as compared to usual care?

Patients with NSCLC will be enrolled in the study from 1 month postoperatively up to 1 year postoperatively. They will be randomized in either the intervention group or the control group.

Patients randomized in the intervention group will be asked to enter a 12-week physical activity telecoaching program with the aim to enhance their physical activity. The telecoaching programs consists of 4 pilars:

1. A wearable (Fitbit) to measure and give feedback on their daily step count.
2. A smartphone coaching application, installed on a smartphone and linked to the wearable, providing automated coaching by displaying an individual activity goal (expressed as daily step count) and daily and weekly feedback on the performance (steps) of the patient.
3. A one-to-one semi-structured interview with the coach discussing the importance of physical activity, motivation, self-efficacy, barriers, favourite activities, and (coping) strategies to become more active resulting in an individual action plan.
4. Phone calls by the coaches initiated in pre-defined situations (non-compliance with wearing the step counter, failure to transmit the data, failure to progress).

Patients randomized in the control group will remain their usual care and will not enter the 12-week physical activity telecoaching program.

DETAILED DESCRIPTION:
Lung cancer is the most commonly diagnosed cancer in men and the third most commonly diagnosed cancer in women worldwide. In Belgium specifically 8874 new cases of lung cancer were diagnosed in 2019 with a poor prognosis (five-year survival rate of 11% to 18%). Non-small cell lung cancer (NSCLC) is the most common subtype of lung cancer, accounting for approximately 85% of all cases. Survival from NSCLC is considerably better than for small-cell lung cancer (SCLC) and depends on the stage of the disease. Complete surgical resection (with or without adjuvant systemic therapy) is the preferred option for patients with resectable (stage I-IIIA) NSCLC.

Existing evidence supports the many benefits, such as blood pressure lowering, higher VO2max levels, lower mortality risk, etc. of physical activity (PA, i.e. all activities that a person performs during a day) among lung cancer survivors. PA however, is proven to be reduced in these patients. A lack of PA can contribute to the perceived symptom burden and decreased health-related quality of life in patients cured from or being treated for NSCLC.

Improving PA is a potential strategy to improve quality of life and symptom experience in these patients. This can possibly be achieved by implementing a (semi-)automated PA tele coaching program to improve PA. The efficacy and effectiveness of implementing such PA tele coaching program for operatively treated NSCLC patients will be assessed in the present study.

A previous study already showed the feasibility and effectiveness of a (semi)-automated tele coaching program (application installed on a smartphone device with real time feedback and motivational messages) and a step counter (Fitbit) providing direct feedback on total daily number of steps, walking time, time in at least moderate PA and movement intensity during walking in patients with chronic obstructive pulmonary disease (COPD).

However, studies investigating the implementation of this application in patients with NSCLC are lacking. Whereas it is clear that research on other populations cannot be generalized to cancer survivors, the investigators are convinced that this previous expertise in COPD can be translated to this population.

Patients who had lung surgery for resectable NSCLC (stage I-IIIA) one to twelve months before inclusion, with or without (neo-)adjuvant chemotherapy/radiotherapy/immunotherapy will be randomized in the intervention group or control group. Patients receiving active immunotherapy following adjuvant chemotherapy can also be included.

The intervention group will receive a 12-week individualized physical activity tele coaching program. Patients randomized in the control group will remain their usual care and will not enter the 12-week physical activity telecoaching program.

After the first 12 weeks, both groups will be followed up for another 12 weeks and also up to 1 year after randomisation.

90 Patients will be included. Patients will be randomised into the intervention or control group. Random blocks of 4 and 6, stratified by adjuvant systemic treatment (yes vs no) and centre of inclusion (Gent, Hasselt) will be used. The upcoming allocation will be concealed using the REDCap randomization module.

The aims of the present study are:

1. Primary objective:

   To investigate the effectiveness and acceptability of a 12-week (semi)automated low-to-moderate intensity PA tele coaching program on physical activity (mean steps per day) in resectable (stage I-IIIA) NSCLC patients after lung surgery, as compared to usual care.
2. Secondary objectives:

A. To investigate the effectiveness of a 12-week (semi)automated low-to-moderate intensity PA tele coaching program on physical activity (MVPA, daily walking time, movement intensity during walking, sedentary time, intensity measured as VMU relative to the VMU during 6MWT), functional exercise capacity, symptoms (dyspnea, fatigue, anxiety), quality of life, quadriceps muscle force and functional performance in resectable (stage I-IIIA) NSCLC patients after lung surgery.

B. To investigate the long-term (24 weeks after randomization) effect of a 12 week (semi)automated low intensity PA tele coaching program on physical activity, functional exercise capacity, symptoms (dyspnea, fatigue, anxiety), quality of life, quadriceps muscle force and functional performance in resectable (stage I-IIIA)NSCLC patients after lung surgery.

C. To explore the intensity of physical activity level relative to the maximal intensity performed during a six minutes walk test and relate this to the improvements in the secondary outcomes.

D.To investigate the association between changes in PA, functional exercise capacity and health-related quality of life (SF-36, EORTC-QLQ-C30, EORTC-QLQ-LC-13) and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Resectable (I-IIIA) NSCLC patients who had lung resection surgery, one to twelve months before inclusion, with or without (neo-)adjuvant chemotherapy/radiotherapy/immunotherapy.
* If patients received adjuvant chemotherapy/radiotherapy, the inclusion window is one months to twelve months after the end of adjuvant chemotherapy/radiotherapy.
* If patients receive adjuvant immunotherapy after the end of adjuvant chemotherapy, patients can be included during the immunotherapy.
* Adults (18+ year)
* Patients who do not systematically perform structured exercise or are planned to do so.
* Ability to give informed consent

Exclusion Criteria:

* Patients having progressive or recurrent lung cancer
* Patients who had other malignancies in the last 2 years
* Psychiatric disorders that preclude them from participation in a physical activity intervention and/or performing the test battery
* Unable to learn to work with a new electronic device (e.g. smartphone)
* Not understanding and speaking Dutch
* Patients with comorbidities or other treatments that preclude them from participation in a physical activity intervention and/or performing the test battery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Mean steps per day | At randomisation, 12 weeks after randomisation
  Change in physical activity (mean steps per day), objectively measured by avalidated tri-axial accelerometer (Dynaport MoveMonitor) after a 12-week(semi)automated low-to-moderate intensity PA tele coaching program. At least 3 valid weekdays (>8 hours of wearing time during the day) is necessary to label this as a valid measurement.

SECONDARY OUTCOMES:
Mean steps per day (measured by Dynaport) | 24 weeks after randomisation, 1 year after the start of the intervention
  Change in physical activity (mean steps per day), objectively measured by avalidated tri-axial accelerometer (Dynaport MoveMonitor) after a 12-week(semi)automated low-to-moderate intensity PA tele coaching program. At least 3valid weekdays (>8 hours of wearing time during the day) is necessary to label this as a valid measurement.
Time in MVPA (moderate-to-vigorous-intense physical activity) | at randomisation, 12 weeks after randomisation, 24 weeks after randomisation, 1 year after the start of the intervention
  Change in time in MVPA, objectively measured by avalidated tri-axial accelerometer (Actigraph) after a 12-week(semi)automated low-to-moderate intensity PA tele coaching program. At least 3valid weekdays (>8 hours of wearing time during the day) is necessary to label thisas a valid measurement.
Walking time | at randomisation, 12 weeks after randomisation, 24 weeks after randomisation, 1 year after the start of the intervention
  Change in walking time, objectively measured by avalidated tri-axial accelerometer (Dynaport Movemonitor) after a 12-week(semi)automated low-to-moderate intensity PA tele coaching program. At least 3 valid weekdays (>8 hours of wearing time during the day) is necessary to label this as a valid measurement.
Movement intensity during walking | at randomisation, 12 weeks after randomisation, 24 weeks after randomisation, 1 year after the start of the intervention
  Change in movement intensity during walking, objectively measured by avalidated tri-axial accelerometer (Dynaport Movemonitor) after a 12-week(semi)automated low-to-moderate intensity PA tele coaching program. At least 3 valid weekdays (>8 hours of wearing time during the day) is necessary to label this as a valid measurement.
Sedentary time | at randomisation, 12 weeks after randomisation, 24 weeks after randomisation, 1 year after the start of the intervention
  Change in sedentary time, objectively measured by avalidated tri-axial accelerometer (Actigraph) after a 12-week(semi)automated low-to-moderate intensity PA tele coaching program. At least 3 valid weekdays (>8 hours of wearing time during the day) is necessary to label this as a valid measurement.
Physical activity intensity measured as VMU (Actigraph) relative to the VMU during 6MWT | AT randomisation, during week 4 and 8 of the intervention and follow-up period, 12 weeks after randomisation, 24 weeks after raondomsation
  A clinically relevant test to measure a patient's exercise capacity is the 6MWT. During this 6MWT the maximal intensity that a patient reaches during the test will be instrumented by the Actigraph. As the maximal intensity we will retrieve the mean VMU during the 6MWT. Day-by-day intensity can then be expressed as a % of this maximum.
Functional exercise capacity measured by 6MWT | At randomisation, 12 weeks after randomisation, 24 weeks after randomisation
  Functional exercise capacity will be measured using a six-minute walk distance (6MWD) test. This test is a routinely used, valid, reliable and safe exercise test in patients with chronic respiratory diseases. The test is standardized in a 30m corridor and will be performed according to the protocol proposed by ERS/ATS.
  Heart rate and oxygen saturation are measured before, during and after the test. Symptom scores for dyspnea and leg fatigue are assessed, at the beginning and end of the test, by the BORG scale. The 6MWD will be measured twice per visit.
Functional exercise capacity measured by 1-min sit-to-stand | At randomisation, 12 weeks after randomisation, 24 weeks after randomisation
  Functional exercise capacity will be measured by a 1-min sit-to-stand (1MSTS) test and is a reliable, valid and responsive test for measuring functional exercise capacity in COPD patients. The 6MWD will be measured twice per visit.
Symptoms of dyspnea | At randomisation, 12 weeks after randomisation, 24 weeks after randomisation; 1 year after the start of the intervention
  The San Diego Shortness of Breath Questionnaire (SOBQ) will be used to assess self-reported shortness of breath while performing activities of daily living. Scores range from 0 (better) to 120 (worse).
Symptoms of fatigue | At randomisation, 12 weeks after randomisation, 24 weeks after randomisation, 1 year after the start of the intervention
  Measured by Functional Assessment of Chronic Illness Treatment-Fatigue (FACIT-F). Maximum score is 160 and minimum score is 0. The higher the score, the better the quality of life.
Symptoms of anxiety, stress and depression | At randomisation, 12 weeks after randomisation, 24 weeks after randomisation, 1 year after the start of the intervention
  Measured by the Depression, Anxiety and Stress scale (short-form) (DASS-21). For each scale it is needed to sum the scores for identified items. Because the DASS-21 is a short form version of the DASS (the long form has 42 items), the final score of each item groups needs to be multiplied by 2.
  Interpretation of Depression score: 0-4=normal, 5-6=mild, 7-10=moderate, 11-13=severe, 14+=extremely severe.
  Interpretation of Anxiety score: 0-3=normal, 4-5=mild, 6-7=moderate, 8-9=severe, 10+=extremely severe.
  Interpretation of Stress score: 0-7=normal, 8-9=mild, 10-12=moderate, 13-16=severe, 17+=extremely severe.
Symptoms of loneliness | At randomisation, 12 weeks after randomisation, 24 weeks after randomisation, 1 year after the start of the intervention
  The UCLA Loneliness Scale provides a reliable and valid assessment of loneliness across a variety of populations and data-collection methods. The total score ranges from 20 to 80. Higher scores indicate higher loneliness. The most commonly used categorization is the following: 20-34 denotes a low degree of loneliness, 35-49 a moderate degree of loneliness, 50-64 a moderately high degree of loneliness, and 65-80 a high degree of loneliness.
Health related quality of life measured by EORTC QLQ-C30-LC13 | At randomisation, 12 weeks after randomisation, 24 weeks after randomisation, 1 year after the start of the intervention
  The European Organization for the Research and Treatment of Cancer Questionnaire and lung cancer module (EORTC QLQ-C30-LC13) is a clinically valid and useful tool for assessing disease- and treatment-specific symptoms in lung cancer patients participating in clinical trials, when combined with the EORTC core quality of life questionnaire. Scores for the EORTC-C30-QLQ and the lung cancer module each range from 0-100. Higher scores indicate a higher quality of life.
General health status measured by SF-36 | At randomisation, 12 weeks after randomisation, 24 weeks after randomisation, 1 year after the start of the intervention
  Measured by the 36-item Short Form Survey (SF-36). SF-36 scores range from 0 (worst) to 100 (best). Higher scores indicate a better quality of life.
General health status measured by EQ-5D-5L | At randomisation, 12 weeks after randomisation, 24 weeks after randomisation, 1 year after the start of the intervention
  The EQ-5D is a short questionnaire to assess general health status. There are 3,125 possible health states defined by combining one level from each dimension, ranging from 11111 (full health) to 55555 (worst health). The instrument also includes a visual analogue scale (EQ-VAS) which provides a single global rating of self-perceived health and is scored on a 0 to 100 mm scale representing "the worst…" and "the best health you can imagine", respectively.
Motivation and self-efficacy measured by Exercise Self-Efficacy Scale (ESES) | At randomisation, 12 weeks after randomisation, 24 weeks after randomisation, 1 year after the start of the intervention
  The Exercise Self-Efficacy Scale (ESES) is a scale developed to measure a person's beliefs or confidence that they can perform various physical activities and exercise on a scale of 1-4. Scores range from 10 (worst) to 40 (best).
Self-efficacy by the modified Tampa Scale for Kinesiophobia (TSK) | At randomisation, 12 weeks after randomisation, 24 weeks after randomisation, 1 year after the start of the intervention
  The modified Tampa Scale for Kinesiophobia (TSK) is a 17-item questionnaire that quantifies fear of movement [32]. Scores range from 17 (best) - 68 (worst).
Self-efficacy measured by Perceived physical activity scale | At randomisation, 12 weeks after randomisation, 24 weeks after randomisation, 1 year after the start of the intervention
  The LIVAS is a questionnaire, tapping how a person perceives his or her physical abilities. The scale is based on the Perceived Physical Ability (PPA) scale (Ryckman et al., 1982). The questionnaire consists of 10 items, asking subjects to evaluate their physical abilities compared to other people of their own age.
  The items have to be rated on a five-point scale.The scale scores therefore vary between 10 and 50. Higher scores represent more positive physical self-efficacy beliefs.
Self-efficacy measured by self-Regulated Questionnaire-Exercise (SRQ-E) | At randomisation, 12 weeks after randomisation, 24 weeks after randomisation, 1 year after the start of the intervention
  The self-Regulated Questionnaire-Exercise (SRQ-E) is a validated 16-item instrument including four regulation subscales used to assesses regulation styles (i.e., intrinsic motivation, identified regulation, introjected regulation and external regulation) in the participants. Using this instrument, participants will be asked reasons for exercising on a regular basis. There are four different types of behavioral regulation. They are external regulation, introjected regulation, identified regulation, and integrated regulation, in order from the least to the most fully internalized. Each participant gets a score on each subscale by averaging responses to each of the items that make up that subscale--for example, the average of all items representing introjected regulation would represent the score for that subscale.
Real time assessment of experience and behaviour | At randomisation, during week 4 and 8 of the intervention and follow-up period, 12 weeks after randomisation, 24 weeks after randomisation, 1 year after the start of the intervention
  Measured by Ecological Momentary Assessment (EMA) measured by m-Path smartphone application
Functional performance | At randomisation, 12 weeks after randomisation, 24 weeks after randomisation
  Measured by the Short Physical Performance Battery (SPPB)This test assesses lower extremity function and mobility. It consists of 3 subtests that are scored and points are added up:
  1. 4-meter gait speed
  2. 5 times sit to stand
  3. Balance test: In this test, patients take specific positions (side by side stand, semi-tandem stand and tandem stand) for a maximum of 10 seconds after demonstration of each foot position. Progressively the foot positions become more difficult.
  Rating of the SPPB: Each task is scored out of 4 (0: worst performance - 4: best performance), with a total score from the tree subtests ranging from 0 (lower level of function) to 12 (higher level of function).
Sleep Quality | At randomisation, during week 4 and 8 of the intervention and follow-up period, 12 weeks after the randomization, 24 weeks after randomization and 1 year after the start of the intervention.
  The Pittsburgh Sleep Quality Index (PSQI) is a self-reported questionnaire assessing sleep quality and patterns over the last month. The questionnaire consists of 19 items, divided into 7 domains: duration of sleep, sleep disturbance, sleep latency, day dysfunction due to sleepiness, sleep efficiency, overall sleep quality, and the need for medications to sleep. The PSQI has a total score between 0 and 21, where higher scores indicate a lower sleep quality. A score of 5 or more often indicates clinically significant sleep problems.

OTHER OUTCOMES:
Time to cancer recurrence | 1 year after the start of the intervention
  by having access to the patients' file for 2years
Time to return to work | up to 2 year after finishing the 12-week intervention
  by having access to the patients' file for 2years
Time to new cancer-related hospital admission | up to 2 year after finishing the 12-week intervention
  by having access to the patients' file for 2years
Need for follow-up cancer treatment. | up to 2 year after finishing the 12-week intervention
  Is there need for follow-up cancer treatment? Will be documented by having access to the patients' file for 2years
Type of follow-up cancer treatment. | up to 2 year after finishing the 12-week intervention
  The type of follow-up cancer treatment will be documented by having access to the patients' file for 2years
Time to death | up to 2 year after finishing the 12-week intervention
  by having access to the patients' file for 2years
Adverse events | up to 2 year after finishing the 12-week intervention
  All adverse events will be collected and graded based on CTCAE 5.0 with information on severity, seriousness, relatedness to the intervention and sequelae; All interactions with the smartphone application and contacts with the coaches will be logged;
Patient experience | 12 weeks after randomisation, 24 weeks after randomisation
  An interview will be performed to ask the patient about their experience of the intervention. The interview is a one-to-one voice-recorded interview with open-ended questions, taken by the researcher.
Patient experience | 12 weeks after randomisation, 24 weeks after randomisation
  A questionnaire will be performed to ask the patient about their experience of the intervention. The questionnaire is on paper and will be filled out by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Stevens, MD, Principal Investigator — University Hospital, Ghent
Locations (6):
- Belgium (6):
  - Ziekenhuis Oost-Limburg, Genk, Limburg
  - Hasselt University, Hasselt, Limburg
  - Jessa Ziekenhuis, Hasselt, Limburg
  - Ghent University Hospital, Ghent, Oost-Vlaanderen
  - AZ Sint-Jan, Bruges, West-Vlaanderen
  - AZ Delta, Roeselare, West-Vlaanderen